CLINICAL TRIAL: NCT01913483
Title: ENDOvascular Interventions With AngioMAX: The ENDOMAX Trial
Acronym: ENDOMAX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDCO-BIV-12-03
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Endovascular Interventions; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bivalirudin (Experimental): Bivalirudin was administered as an intravenous (IV) bolus and infusion for the duration of the procedure (mean duration of 48.6 minutes). The bolus (0.75 milligrams (mg)/kilogram [kg]) was administered via systemic IV administration. Immediately after the bolus, an IV infusion of bivalirudin was initiated at a dose of 1.75 mg/kg/hour (h) (or 1 mg/kg/h for participants with an estimated glomerular filtration rate [eGFR] <30 milliliters/minute [mL/min]).
  Interventions: Drug: Bivalirudin
- Unfractionated Heparin (Active Comparator): UFH was administered as an IV bolus for the duration of the procedure (mean duration of 48.6 minutes). UFH was administered via weight-based IV bolus at a dose of 50 units (U)/kg to 70 U/kg. Additional bolus doses were administered per standard-of-care use.
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: Bivalirudin — Bivalirudin is an anticoagulant that binds directly to thrombin in a bivalent and reversible fashion.
  Other Names: AngioMAX; Angiox
  Arms: Bivalirudin
Drug: Unfractionated Heparin — Unfractionated heparin is an anticoagulant.
  Other Names: Heparin
  Arms: Unfractionated Heparin

SUMMARY:
The primary objective of the study is to test whether anticoagulation with bivalirudin results in fewer major bleeding complications compared with unfractionated heparin (UFH) in participants undergoing peripheral endovascular interventions (PEI). The secondary objective is to test whether there were potential benefits from bivalirudin therapy on other clinically important events such as death, myocardial infarction (MI), stroke and/or transient ischemic attack (TIA), amputation, unplanned repeat revascularization (URV), and minor bleeding, as well as potential economic benefits that may result from improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age
* Must be undergoing one of the following PEI procedures:

  * Carotid artery stenting
  * Lower Extremity Interventions (LEI) for Critical Limb Ischemia
  * LEI for claudication
* Provide written informed consent prior to any study-specific procedure being performed

Exclusion Criteria:

* Any known contra-indication to the use of bivalirudin or UFH
* Acute limb ischemia
* Planned amputation regardless of the outcome of the PEI
* Dialysis dependent
* Weight less than 38 kg or more than 202 kg
* History of any bleeding diathesis or severe hematological disease
* History of intra-cranial: mass, aneurysm, arteriovenous malformation or hemorrhage
* Gastrointestinal or genitourinary bleeding within the 30 days prior to randomization
* Any surgery (excluding punch or shave skin biopsy) within the 30 days prior to randomization
* Concomitant percutaneous coronary intervention
* Any percutaneous coronary, endovascular, or structural heart disease procedure within 30 days prior to randomization
* International normalized ratio >1.7 within 24 h prior to the index procedure
* Administration of therapeutic doses of UFH within 30 min prior to the index procedure (a low dose [≤2000 U] of heparin is permitted during the diagnostic angiogram prior to the intervention)
* Administration of enoxaparin within 8 h; other low molecular weight heparins or fondaparinux within 24 h; any oral anti-Xa or antithrombin agent within 48 h; or thrombolytics, glycoprotein inhibitors, or warfarin within 72 h prior to the index procedure
* Severe contrast allergy that cannot be pre-medicated
* Procedures performed by radial access when they are intended as the primary access site for the index procedure
* Known or suspected pregnant women or nursing mothers
* Previous enrollment in this study (MDCO-BIV-12-03)
* Participation in other investigational drug or device trials within 30 days prior to randomization
* Participants who, for any reason, are deemed by the investigator to be inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Tri-Lakes Research, Hot Springs, Arkansas
  - Stanford Hospital and Clinics, Stanford, California
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Florida Research Network, Gainesville, Florida
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Peoria Radiology Research & Education Foundation, Peoria, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Kentucky Heart Foundation - King's Daughters Medical Center, Ashland, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - VA Boston Healthcare System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Michigan Heart, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Integris - Baptist Medical Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Tech University Health Science Center, Lubbock, Texas
  - Scott and White Hospital, Temple, Texas
  - Alpine Research, Ogden, Utah
  - INOVA Alexandria Hospital, Alexandria, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were randomized into the trial, who received at least one dose of study drug (Safety Population), and underwent the index peripheral endovascular interventions (PEI) procedure were included in the modified Intent-to-Treat (mITT) Population. This was the primary population for analyses of the primary and secondary endpoints.
Groups:
- Bivalirudin: Bivalirudin was administered as an intravenous (IV) bolus and infusion for the duration of the procedure (mean duration of 48.6 minutes). The bolus (0.75 milligrams (mg)/kilogram [kg]) was administered via systemic IV administration. Immediately after the bolus, an IV infusion of bivalirudin was initiated at a dose of 1.75 mg/kg/hour (h) (or 1 mg/kg/h for participants with an estimated glomerular filtration rate [eGFR] <30 milliliters per minute [mL/min]).
- Unfractionated Heparin: Unfractionated heparin (UFH) was administered as an IV bolus for the duration of the procedure (mean duration of 48.6 minutes). UFH was administered via weight-based IV bolus at a dose of 50 units (U)/kg to 70 U/kg. Additional bolus doses were administered per standard-of-care use.
Period: Overall Study
Arm/Group | Bivalirudin | Unfractionated Heparin
Started (All participants who were randomized to the study were included in the Intent-to-Treat Population.) | 367 | 365
Received at Least 1 Dose of Study Drug (The 656 participants were the same participants for both the Safety Population and mITT Population.) | 335 | 321
Completed (One participant in the Bivalirudin and UFH Arms each died before receiving study drug.) | 346 | 343
Not Completed | 21 | 22
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 6 | 3
Not completed — Death | 14 | 17

BASELINE CHARACTERISTICS:
Population: mITT Population: Participants who were randomized into the trial, received at least one dose of study drug, and underwent the index PEI procedure.
Groups:
- Bivalirudin: Bivalirudin was administered as an IV bolus and infusion for the duration of the procedure (mean duration of 48.6 minutes). The bolus (0.75 mg/kg) was administered via systemic IV administration. Immediately after the bolus, an IV infusion of bivalirudin was initiated at a dose of 1.75 mg/kg/h (or 1 mg/kg/h for participants with an eGFR <30 mL/min).
- Unfractionated Heparin: UFH was administered as an IV bolus for the duration of the procedure (mean duration of 48.6 minutes). UFH was administered via weight-based IV bolus at a dose of 50 U/kg to 70 U/kg. Additional bolus doses were administered per standard-of-care use.
- Total: Total of all reporting groups
Arm/Group | Bivalirudin | Unfractionated Heparin | Total
Number analyzed (Participants) | 335 | 321 | 656
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (10.3) | 68.8 (10.3) | 69.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 123 | 256
  Male | 202 | 198 | 400
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 40 | 89
  White | 282 | 278 | 560
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 335 | 321 | 656

OUTCOME MEASURES:

1. Primary Outcome: Participants With Bleeding Academic Research Consortium Type 3 or Greater (BARC ≥3) Events Up to 48 h or at Hospital Discharge, As Adjudicated by the Independent Clinical Events Committee (CEC)
Description: BARC ≥3 includes:
  Type 3a-3c: clinical, laboratory, and/or imaging evidence of bleeding, which includes any transfusion with overt bleeding, bleeds that result in surgical intervention or administration of IV vasoactive drugs, overt bleeds with a hemoglobin drop greater than or equal to 3 grams (g)/deciliters (dL) to greater than or equal to 5 g/dL, cardiac tamponade caused by bleeding, intracranial hemorrhage, and intraocular bleeds that compromise vision.
  Type 4: (Coronary Artery Bypass Grafting-related Bleeding) includes perioperative intracranial bleeding within 48 h, bleeds that result in reoperation following closure of sternotomy for the purpose of controlling bleeding, bleeds that result in treatment with transfusion of ≥5 U of whole blood or packed red blood cells within a 48-h period; and chest tube output ≥2 liters within a 24-h period.
  Type 5: fatal bleeding that directly results in death that is either clinically suspicious or is confirmed as the cause of death.
Time Frame: Study drug administration (Day 1) up to 48 h post study drug initiation or at hospital discharge, whichever occurs first
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin
Number analyzed (Participants) | 335 | 321
percentage of participants | 1.5 | 1.6
Statistical Analysis 1: Comparison: Bivalirudin vs Unfractionated Heparin; Assuming a bleeding event rate of 5.0% in the heparin control treatment group and 3.2% in the bivalirudin group (36% relative risk reduction, a sample size of 3900 participants was to provide more than 80% power with a two-tailed alpha level of 0.05). This estimate took into consideration that the interim efficacy analysis was to be performed when approximately 70% of participants were enrolled using the O'Brien-Fleming alpha spending function; Test type: Superiority; p = 0.9458, Chi-squared — The primary endpoint analysis was to assess the superiority of bivalirudin versus UFH in BARC ≥3 bleeds within the 48 hours post study drug initiation or at hospital discharge, whichever occurred first

2. Secondary Outcome: Participants With Myocardial Infarction (MI), Stroke/Transient Ischemic Attack (TIA), Unplanned Repeat Revascularization (URV), Death, and Minor Bleeding Up to 48 h Post Study Drug Administration
Description: Outcome assessments at 48 h post study drug initiation include bleeding events defined as BARC Type 2 or greater (BARC ≥2), bleeding events defined as thrombolysis in myocardial infarction (TIMI) major and TIMI minor, and net adverse clinical events (NACE) as adjudicated by the CEC (NACE=death, MI, stroke/TIA, amputations, URV, or bleeding events defined as BARC ≥3).
  In addition to Type 3(a-c), 4, and 5, BARC ≥2 also includes Type 2 bleeding, which is any overt, actionable sign of hemorrhage (more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for Type 3, 4, or 5, but does meet at least one of the following criteria of: requiring nonsurgical, medical intervention by a health-care professional; leading to hospitalization or increased level of care; prompting evaluation.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Bivalirudin | Unfractionated Heparin
Number analyzed (Participants) | 335 | 321
participants
  Bleed (BARC ≥ Type 2) | 47 | 42
  TIMI major | 0 | 4
  TIMI minor | 4 | 1
  Death | 0 | 1
  MI | 0 | 0
  Stroke/TIA | 0 | 0
  Amputation | 0 | 0
  URV | 2 | 2
  NACE | 7 | 6

3. Secondary Outcome: Participants With MI, Stroke/TIA, URV, Death, or Minor Bleeding Up to Day 30
Description: Outcome assessments at Day 30 include NACE, Major Adverse Clinical Events (MACE=death, MI, stroke/TIA, amputation, or URV), and bleeding defined as BARC ≥2, as adjudicated by the CEC.
  In addition to Type 3(a-c), 4, and 5, BARC ≥2 also includes Type 2 bleeding, which is any overt, actionable sign of hemorrhage (more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for Type 3, 4, or 5, but does meet at least one of the following criteria of: requiring nonsurgical, medical intervention by a health-care professional; leading to hospitalization or increased level of care; prompting evaluation.
Time Frame: Study drug initiation (Day 1) up to 30 days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Bivalirudin | Unfractionated Heparin
Number analyzed (Participants) | 335 | 321
participants
  Bleed (BARC ≥ Type 2) | 53 | 51
  Bleed (BARC ≥ Type 3) | 6 | 7
  Death | 2 | 3
  MI | 0 | 1
  Stroke/TIA | 1 | 2
  Amputation | 8 | 5
  URV | 9 | 11
  MACE (Death/MI/Stroke/Amputation/URV) | 18 | 19
  NACE | 22 | 23

ADVERSE EVENTS:
Time Frame: Randomization up to 30 days (±7 days)
Description: Does not include 2 participants who died before receiving study drug.
Arm/Group | Bivalirudin | Unfractionated Heparin
All-Cause Mortality (participants affected / at risk) | 13/335 | 16/321
Serious Adverse Events (participants affected / at risk) | 25/335 | 27/321
Other Adverse Events (participants affected / at risk) | 81/335 | 70/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bivalirudin (N=335) | Unfractionated Heparin (N=321)
Cellulitis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 3
Postoperative wound infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 2 | 0
Groin infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Femoral artery dissection (Vascular disorders) | 0 | 1
Femoral artery embolism (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral artery dissection (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Ischaemic ulcer (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 0 | 1
Vessel puncture site pain (General disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Surgical and medical procedures) | 0 | 1
Peripheral artery bypass (Surgical and medical procedures) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Mental status change (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bivalirudin (N=335) | Unfractionated Heparin (N=321)
Hypertension (Vascular disorders) | 15 | 13
Hypotension (Vascular disorders) | 10 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8
Groin pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Vessel puncture site pain (General disorders) | 9 | 5
Pain (General disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 8 | 5
Vomiting (Gastrointestinal disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No